CLINICAL TRIAL: NCT05666206
Title: Efficacy of Fibrin Sealant in Hypospadias Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibrin sealant in hypospadius
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrin group (Active Comparator): Fibrin sealant covered with 2ry dartos flap.
  Interventions: Procedure: fibrin sealant in hypospadias
- Standard TIP technique (Active Comparator): standard TIP technique with second dartos flap and no use of fibrin sealant
  Interventions: Procedure: fibrin sealant in hypospadias

INTERVENTIONS:
Procedure: fibrin sealant in hypospadias — fibrin sealant will be used over the suture line

SUMMARY:
The aim of the study was to evaluate if application of a fibrin sealant over the urethroplasty suture line for waterproofing instead of a dartos vascularized pedicled flap to reduce complications and improve the outcome in hypospadias repair.

DETAILED DESCRIPTION:
Many procedures have been tried for the sake of proper management of hypospadias and reducing the complications. Of them, tabularized incised plate (TIP) is one of the most convenient technique, which became the most common procedure for hypospadias repair (Elsayem et al., 2022).

Although many surgical modifications and techniques have been prescribed to minimize post-operative complications and improve outcomes, a high percentage of complications still occurs. Urethrocutaneous fistulae are the most common post-operative complication (10%-40%) after hypospadias surgery; other complications being skin flap related complications such as flap necrosis, suture line breakdown, ascent of the testis and penile torsion (Shenoy et al.,2021).

In this thesis a secondary preputial dartos flap will be performed in all cases and we will evaluate the value of usage of fibrin glue on the 1ry suture line .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria All treatment naïve children with hypospadias.

Exclusion Criteria:

* Adult hypospadias.
* Recurrent cases.
* Prio pelvic trauma or radiation.

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Success of surgery | 3 months
  Number of patients with good stream, normal looking meatus and no need for auxiliary maneuvers.

SECONDARY OUTCOMES:
complications of hypospadias surgery | 3 months
  Number of patients with fistula, chordee, rotation, ....

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided